CLINICAL TRIAL: NCT03089879
Title: A Phase 1, Open Label, Non-randomized, Single Center Study to Evaluate the Safety and Immunogenicity of 1 Booster Vaccination With (GVGH Shigella Sonnei 1790GAHB) Vaccine Administered Intramuscularly in Healthy Adults Previously Primed With Three Doses of the Same Vaccine in Study H03_01TP Compared to 1 Vaccination With (1790GAHB) Administered Intramuscularly Either to Subjects Who Received Placebo in the H03_01TP Study or naïve Subjects Who Were Not Part of H03_01TP Study
Brief Title: A Study to Evaluate Safety and Immunogenicity of 1 Booster Dose of 1790GAHB Vaccine in Healthy Adults Primed With 3 Doses of 1790GAHB Vaccine in Study H03_01TP Compared to 1 Vaccination of 1790GAHB in Either Subjects Who Received Placebo in the Same Study or naïve Subjects Not Part of H03_01TP Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 205905; 2016-004178-16 (EudraCT Number)
Record Dates: First submitted 2017-03-21; First posted 2017-03-24 (Actual); Results first posted 2019-03-07 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Dysentery, Bacillary
Keywords: Immunogenicity, Vaccine; Immunologic Memory; GMMA; Shigella Vaccines; Shigellosis; Dysentery, Bacillary; Healthy Volunteers; Safety; Bacteria; Clinical Trials, Phase 1; Shigella sonnei
MeSH Terms: conditions — Dysentery, Bacillary

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Shigella Group (Experimental): Healthy male and female subjects, aged 22 to 50 years, previously primed with 3 doses of the GVGH Shigella sonnei 1790GAHB vaccine in the H03_01TP parent study and who had undetectable antibody titers at baseline, received one intramuscular booster dose of the same vaccine in the current study, at Day 1.
  Interventions: Biological: GVGH Shigella sonnei 1790GAHB vaccine
- Placebo Group (Experimental): Healthy male and female subjects, aged 22 to 50 years, who previously received placebo in the H03_01TP parent study and who had undetectable antibodies at baseline, received one intramuscular GVGH Shigella sonnei 1790GAHB vaccine dose in the current study, at Day 1.
  Interventions: Biological: GVGH Shigella sonnei 1790GAHB vaccine
- Naïve Group (Experimental): Healthy male and female subjects, aged 22 to 50 years, who were not part of H03_01TP parent study, received one intramuscular GVGH Shigella sonnei 1790GAHB vaccine dose in the current study, at Day 1.
  Interventions: Biological: GVGH Shigella sonnei 1790GAHB vaccine

INTERVENTIONS:
Biological: GVGH Shigella sonnei 1790GAHB vaccine — Single dose administered at Day 1, by intramuscular injection.

SUMMARY:
GVGH Shigella Sonnei 1970GAHB is a vaccine aimed at preventing the disease caused by Shigella sonnei.

A post-hoc analysis of subjects who participated in the parent study showed significantly different responses in subjects with detectable versus undetectable antibody titres at baseline, suggesting the possibility that the vaccine might not be sufficiently immunogenic in completely naïve adults.

This study was then designed to further characterize the immunogenicity profile of the vaccine and to evaluate whether it was able to induce an immunological memory response.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, aged 22 to 50 years, who were previously vaccinated, with either vaccine (3 doses) or placebo, in H03_01TP and who had undetectable antibody titers at baseline, or Males and females, aged 22 to 50 years, who were not part of H03_01TP.
* Individuals who, after the nature of the study has been explained to them, and prior to any protocol specific procedures being performed, have given written consent according to local regulatory requirements.
* Individuals in good health as determined by the outcome of medical history, physical examination, hematological blood tests and clinical judgment of the investigator.
* If women of child-bearing potential, have a negative urinary pregnancy test prior study vaccination and willingness to use acceptable birth control measures for the entire study duration.
* Individuals affiliated to a social security regimen.

Exclusion Criteria:

* Individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the subject's ability to participate in the study.
* Individuals with any progressive or severe neurological disorder, seizure disorder or Guillain-Barré syndrome.
* Individuals who are not able to understand and to follow all required study procedures for the whole period of the study.
* Individuals with known hepatitis B or C or suspected HIV infection or HIV related disease with history of an autoimmune disorder or any other known or suspected impairment /alteration of the immune system.
* Progressive, unstable or uncontrolled clinical conditions.
* Hypersensitivity, including allergy, to any component of vaccines, medicinal products or medical equipment whose use is foreseen in this study.
* Individuals with a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
* Clinical conditions representing a contraindication to intramuscular vaccination and blood draws.
* Abnormal function of the immune system resulting from:

  * Clinical conditions;
  * Systemic administration of corticosteroids for more than 14 consecutive days within 90 days prior to informed consent;
* Administration of antineoplastic and immunomodulating agents or radiotherapy within 90 days prior to informed consent.
* Received immunoglobulins or any blood products within 180 days prior to informed consent.
* Study personnel as an immediate family or household member.
* Any other clinical condition that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subject due to participation in the study.
* Individuals who have received an investigational product in another clinical trial 28 days prior to first study visit or intent to receive another investigational product at any time during the conduct of this study.
* Individuals who received any other vaccines within 4 weeks prior to enrollment in this study or who are planning to receive any vaccine within the entire study duration. Inactivated influenza vaccine can be given, but only 4 weeks earlier or 4 weeks later than the date of immunization.
* Individuals who have received blood, blood products, and/or plasma derivatives including parenteral immunoglobulin preparations in the past 180 days.
* Individuals with body temperature > 38.0 degrees Celsius within 3 days of intended study vaccination.
* Individuals with Body Mass Index > 30 kg/m2.
* Individuals with history of substance or alcohol abuse within the past 2 years.
* Women who are pregnant or are breast-feeding, or are of childbearing age who have not used or do not plan to use acceptable birth control measures, for the duration of the study.
* Females with history of stillbirth, neonatal loss, or previous infant with anomaly.
* Individuals who have a previously laboratory confirmed or suspected disease caused by S. sonnei.
* Individuals who have had household contact with/and or intimate exposure to an individual with laboratory confirmed S. sonnei.
* Any condition, which, in the opinion of the investigator may pose an increased and unreasonable safety risk to the subject if participating to the present study.
* Individuals with a neutrophil count value lower than 1.8 10^9/L at screening assessment.
* Individuals with human leukocyte antigen (HLA)-B27 positive and/or with history of reactive arthritis.
* Previous history of Benign Ethnic Neutropenia or drug related Neutropenia and/or concomitant treatment with neutropenic agents.

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/SearchAllPostings.aspx?searchparam=200147

REFERENCES:
- [Background] Launay O, Ndiaye AGW, Conti V, Loulergue P, Scire AS, Landre AM, Ferruzzi P, Nedjaai N, Schutte LD, Auerbach J, Marchetti E, Saul A, Martin LB, Podda A. Booster Vaccination With GVGH Shigella sonnei 1790GAHB GMMA Vaccine Compared to Single Vaccination in Unvaccinated Healthy European Adults: Results From a Phase 1 Clinical Trial. Front Immunol. 2019 Mar 8;10:335. doi: 10.3389/fimmu.2019.00335. eCollection 2019. PMID 30906291
- [Derived] Micoli F, Rossi O, Conti V, Launay O, Scire AS, Aruta MG, Nakakana UN, Marchetti E, Rappuoli R, Saul A, Martin LB, Necchi F, Podda A. Antibodies Elicited by the Shigella sonnei GMMA Vaccine in Adults Trigger Complement-Mediated Serum Bactericidal Activity: Results From a Phase 1 Dose Escalation Trial Followed by a Booster Extension. Front Immunol. 2021 May 4;12:671325. doi: 10.3389/fimmu.2021.671325. eCollection 2021. PMID 34017343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 35 subjects were enrolled into the study. Of these, 7 and 2 eligible subjects from the H03_01TP parent study were enrolled into the Shigella Group and Placebo Group, respectively. 26 subjects were enrolled into the Naïve Group. All 35 subjects were vaccinated and analyzed for immunogenicity and safety.
Pre-assignment Details: The subjects in Naive Group, who were not part of the H03_01TP study, were added in order to have a more balanced number of previously unvaccinated and vaccinated subjects in the extension trial.
Period: Overall Study
Arm/Group | Shigella Group | Placebo Group | Naïve Group
Started | 7 | 2 | 26
Completed | 7 | 2 | 26
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Shigella Group | Placebo Group | Naïve Group | Total
Number analyzed (Participants) | 7 | 2 | 26 | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.7 (7.89) | 40.5 (10.61) | 33.8 (8.41) | 34.9 (8.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 9 | 15
  Male | 3 | 0 | 17 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 0 | 1 | 2
  White | 6 | 2 | 24 | 32
  Unspecified | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Concentrations of Immunoglobulin (IgG) Against Lipopolysaccharide (LPS) S. Sonnei O-antigen
Description: IgG concentrations are expressed as Geometric Mean Concentrations (GMCs), as determined by the Enzyme-linked immunosorbent assay (ELISA) with Shigella sonnei (S.sonnei) O-antigen containing Lipopolysaccharide (LPS) coating antigen. Concentrations are presented as GMCs expressed in ELISA units per milliliter (EU/mL).
Time Frame: At Day 8 (7 days after vaccination)
Population: The analysis was performed on the Full Analysis Set, which included all enrolled subjects who received a study vaccination and provided immunogenicity data at relevant time points.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Shigella Group | Placebo Group | Naïve Group
Number analyzed (Participants) | 7 | 2 | 23
EU/mL | 168 [32 to 889] | 5.17 [0.033 to 810] | 38 [20 to 72]

2. Secondary Outcome: Number of Subjects With Abnormal Haematological Test Values
Description: Assessed haematological parameters are: basophils (BAS), eosinophils (EOS), erythrocytes (ERCS), hematocrit (HCT), hemoglobin (HGB), leukocytes (LKCS), lymphocytes (LYM), monocytes (MONO), neutrophils (NEU) and platelet (PLT).
Time Frame: At Day 8 (7 days after vaccination) and Day 85 (84 days after vaccination)
Population: The analysis was performed on the Overall Safety Set, which included all enrolled subjects who received a study vaccination and for whom solicited and unsolicited adverse event data were available. For the purpose of this analysis, the subjects from Placebo and Naïve Groups were pooled into a single group (Placebo + Naïve Group).
Measure: Count of Participants; unit: Participants
Groups:
- Placebo + Naïve Group: Healthy male and female subjects, aged 22 to 50 years, who previously received placebo in the H03_01TP parent study and who had undetectable antibodies at baseline (Placebo Group), or subjects who were not part of H03_01TP parent study (Naïve Group) were pooled into the Placebo + Naïve Group. All subjects received one intramuscular GVGH Shigella sonnei 1790GAHB vaccine dose in the current study, at Day 1.
Arm/Group | Shigella Group | Placebo + Naïve Group
Number analyzed (Participants) | 7 | 28
Participants
  BAS, Below (baseline) - Within (Day 8) | 0 | 0
  BAS, Within (baseline) - Within (Day 8) | 7 | 28
  BAS, Above (baseline) - Within (Day 8) | 0 | 0
  BAS, Below (baseline) - Within (Day 85) | 0 | 0
  BAS, Within (baseline) - Within (Day 85) | 7 | 28
  BAS, Above (baseline) - Within (Day 85) | 0 | 0
  EOS, Below (baseline) - Below (Day 8) | 1 | 2
  EOS, Within (baseline) - Below (Day 8) | 0 | 1
  EOS, Above (baseline) - Below (Day 8) | 0 | 0
  EOS, Below (baseline) - Within (Day 8) | 1 | 3
  EOS, Within (baseline) - Within (Day 8) | 5 | 21
  EOS, Above (baseline) - Within (Day 8) | 0 | 1
  EOS, Below (baseline) - Below (Day 85) | 1 | 1
  EOS, Within (baseline) - Below (Day 85) | 0 | 0
  EOS, Above (baseline) - Below (Day 85) | 0 | 0
  EOS, Below (baseline) - Within (Day 85) | 1 | 4
  EOS, Within (baseline) - Within (Day 85) | 4 | 22
  EOS, Above (baseline) - Within (Day 85) | 0 | 0
  EOS, Below (baseline) - Above (Day 85) | 0 | 0
  EOS, Within (baseline) - Above (Day 85) | 1 | 0
  EOS, Above (baseline) - Above (Day 85) | 0 | 1
  ERCS, Below (baseline) - Below (Day 8) | 0 | 1
  ERCS, Within (baseline) - Below (Day 8) | 1 | 1
  ERCS, Above (baseline) - Below (Day 8) | 0 | 0
  ERCS, Below (baseline) - Within (Day 8) | 0 | 0
  ERCS, Within (baseline) - Within (Day 8) | 6 | 26
  ERCS, Above (baseline) - Within (Day 8) | 0 | 0
  ERCS, Below (baseline) - Below (Day 85) | 0 | 1
  ERCS, Within (baseline) - Below (Day 85) | 2 | 0
  ERCS, Above (baseline) - Below (Day 85) | 0 | 0
  ERCS, Below (baseline) - Within (Day 85) | 0 | 0
  ERCS, Within (baseline) - Within (Day 85) | 5 | 27
  ERCS, Above (baseline) - Within (Day 85) | 0 | 0
  HCT, Below (baseline) - Below (Day 8) | 2 | 1
  HCT, Within (baseline) - Below (Day 8) | 0 | 0
  HCT, Above (baseline) - Below (Day 8) | 0 | 0
  HCT, Below (baseline) - Within (Day 8) | 0 | 1
  HCT, Within (baseline) - Within (Day 8) | 5 | 26
  HCT, Above (baseline) - Within (Day 8) | 0 | 0
  HCT, Below (baseline) - Below (Day 85) | 2 | 2
  HCT, Within (baseline) - Below (Day 85) | 1 | 0
  HCT, Above (baseline) - Below (Day 85) | 0 | 0
  HCT, Below (baseline) - Within (Day 85) | 0 | 0
  HCT, Within (baseline) - Within (Day 85) | 4 | 26
  HCT, Above (baseline) - Within (Day 85) | 0 | 0
  HGB, Below (baseline) - Below (Day 8) | 2 | 1
  HGB, Within (baseline) - Below (Day 8) | 0 | 0
  HGB, Above (baseline) - Below (Day 8) | 0 | 0
  HGB, Below (baseline) - Within (Day 8) | 0 | 0
  HGB, Within (baseline) - Within (Day 8) | 5 | 27
  HGB, Above (baseline) - Within (Day 8) | 0 | 0
  HGB, Below (baseline) - Below (Day 85) | 2 | 1
  HGB, Within (baseline) - Below (Day 85) | 1 | 1
  HGB, Above (baseline) - Below (Day 85) | 0 | 0
  HGB, Below (baseline) - Within (Day 85) | 0 | 0
  HGB, Within (baseline) - Within (Day 85) | 4 | 26
  HGB, Above (baseline) - Within (Day 85) | 0 | 0
  LKCS, Below (baseline) - Below (Day 8) | 1 | 0
  LKCS, Within (baseline) - Below (Day 8) | 0 | 2
  LKCS, Above (baseline) - Below (Day 8) | 0 | 0
  LKCS, Below (baseline) - Within (Day 8) | 0 | 0
  LKCS, Within (baseline) - Within (Day 8) | 6 | 25
  LKCS, Above (baseline) - Within (Day 8) | 0 | 0
  LKCS, Below (baseline) - Above (Day 8) | 0 | 0
  LKCS, Within (baseline) - Above (Day 8) | 0 | 1
  LKCS, Above (baseline) - Above (Day 8) | 0 | 0
  LKCS, Below (baseline) - Below (Day 85) | 1 | 0
  LKCS, Within (baseline) - Below (Day 85) | 0 | 1
  LKCS, Above (baseline) - Below (Day 85) | 0 | 0
  LKCS, Below (baseline) - Within (Day 85) | 0 | 0
  LKCS, Within (baseline) - Within (Day 85) | 6 | 26
  LKCS, Above (baseline) - Within (Day 85) | 0 | 0
  LKCS, Below (baseline) - Above (Day 85) | 0 | 0
  LKCS, Within (baseline) - Above (Day 85) | 0 | 1
  LKCS, Above (baseline) - Above (Day 85) | 0 | 0
  LYM, Below (baseline) - Below (Day 8) | 2 | 3
  LYM, Within (baseline) - Below (Day 8) | 0 | 1
  LYM, Above (baseline) - Below (Day 8) | 0 | 0
  LYM, Below (baseline) - Within (Day 8) | 0 | 3
  LYM, Within (baseline) - Within (Day 8) | 5 | 21
  LYM, Above (baseline) - Within (Day 8) | 0 | 0
  LYM, Below (baseline) - Below (Day 85) | 1 | 2
  LYM, Within (baseline) - Below (Day 85) | 0 | 2
  LYM, Above (baseline) - Below (Day 85) | 0 | 0
  LYM, Below (baseline) - Within (Day 85) | 1 | 4
  LYM, Within (baseline) - Within (Day 85) | 5 | 20
  LYM, Above (baseline) - Within (Day 85) | 0 | 0
  MONO, Below (baseline) - Within (Day 8) | 0 | 0
  MONO, Within (baseline) - Within (Day 8) | 7 | 28
  MONO, Above (baseline) - Within (Day 8) | 0 | 0
  MONO, Below (baseline) - Within (Day 85) | 0 | 0
  MONO, Within (baseline) - Within (Day 85) | 7 | 28
  MONO, Above (baseline) - Within (Day 85) | 0 | 0
  NEU, Below (baseline) - Within (Day 8) | 0 | 0
  NEU, Within (baseline) - Within (Day 8) | 7 | 28
  NEU, Above (baseline) - Within (Day 8) | 0 | 0
  NEU, Below (baseline) - Within (Day 85) | 0 | 0
  NEU, Within (baseline) - Within (Day 85) | 7 | 28
  NEU, Above (baseline) - Within (Day 85) | 0 | 0
  PLT, Below (baseline) - Within (Day 8) | 0 | 0
  PLT, Within (baseline) - Within (Day 8) | 7 | 28
  PLT, Above (baseline) - Within (Day 8) | 0 | 0
  PLT, Below (baseline) - Within (Day 85) | 0 | 0
  PLT, Within (baseline) - Within (Day 85) | 7 | 28
  PLT, Above (baseline) - Within (Day 85) | 0 | 0

3. Secondary Outcome: Number of Subjects With Solicited Local Adverse Events
Description: Assessed solicited local adverse events include injection site erythema, injection site induration and injection site pain. Any symptom = occurrence of the symptom regardless of intensity grade.
Time Frame: From 30 minutes through Day 7 post-vaccination
Population: The analysis was performed on the Solicited Safety Set, which included all enrolled subjects who received a study vaccination and for whom solicited adverse event data were available. For the purpose of this analysis, the subjects from Placebo and Naïve Groups were pooled into a single group (Placebo+Naïve Group).
Measure: Count of Participants; unit: Participants
Arm/Group | Shigella Group | Placebo + Naïve Group
Number analyzed (Participants) | 7 | 28
Participants
  Any Erythema | 1 | 0
  Any Induration | 0 | 1
  Any Pain | 6 | 24

4. Secondary Outcome: Number of Subjects With Solicited Systemic Adverse Events
Description: Assessed solicited systemic adverse events include arthralgia, chills, fatigue, headache, malaise, myalgia and oral fever. Other indicators of solicited adverse events include prevention of pain and/or fever and treatment of pain and/or fever. Any symptom = occurrence of the symptom regardless of intensity grade. Fever = body temperature (measured orally) equal to or above (≥) 38.0 °C.
Time Frame: From 30 minutes through Day 7 post-vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Shigella Group | Placebo + Naïve Group
Number analyzed (Participants) | 7 | 28
Participants
  Any Arthralgia | 1 | 3
  Any Chills | 1 | 1
  Any Fatigue | 3 | 11
  Any Headache | 1 | 5
  Any Malaise | 1 | 2
  Any Myalgia | 2 | 8
  Fever | 0 | 0
  Prevention of Pain and/or Fever | 0 | 0
  Treatment of Pain and/or Fever | 3 | 5

5. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events
Description: An unsolicited adverse event (AE) is an adverse event that was not solicited using a Subject Diary and that was spontaneously communicated by a subject who has signed the informed consent. Potential unsolicited AEs may be medically attended (defined as symptoms or illnesses requiring hospitalization, or emergency room visit, or visit to/by a health care provider), or were of concern to the subject. Any = occurrence of the symptom regardless of intensity grade. Grade 3 AE = AE that prevented daily activity. Possibly/probably related AE = AE determined by the investigator as possibly related (the administration of the investigational vaccine and AE are considered reasonably related in time and the AE could be explained by exposure to the investigational vaccine or by other causes) or probably related (exposure to the investigational vaccine and AE are reasonably related in time and no alternative explanation has been identified) to the study vaccination.
Time Frame: Throughout the study period (From Day 1 up to Day 85)
Population: The analysis was performed on the Unsolicited Safety Set, which included all enrolled subjects who received a study vaccination and for whom unsolicited adverse event data were available. For the purpose of this analysis, the subjects from Placebo and Naïve Groups were pooled into a single group (Placebo+Naïve Group).
Measure: Count of Participants; unit: Participants
Arm/Group | Shigella Group | Placebo + Naïve Group
Number analyzed (Participants) | 7 | 28
Participants
  Any AE(s) | 4 | 7
  Grade 3 AE(s) | 0 | 0
  Possibly/probably related AE(s) | 0 | 1

6. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: A serious adverse event is defined as an untoward medical occurrence that at any dose resulted in death, was life-threatening, required hospitalization or prolonged hospitalization, resulted in persistent or significant disability/incapacity, or in a congenital anomaly/birth defect; an important and significant medical event that may not be immediately life-threatening or resulting in death or hospitalization but, based upon appropriate medical judgment, may jeopardize the subject or may require intervention to prevent one of the other outcomes listed above.
Time Frame: Throughout the study period (from Day 1 up to Day 85)
Population: The analysis was performed on the Overall Safety Set, which included all enrolled subjects who received a study vaccination and for whom solicited and unsolicited adverse event data were available. For the purpose of this analysis, the subjects from Placebo and Naïve Groups were pooled into a single group (Placebo+Naïve Group).
Measure: Count of Participants; unit: Participants
Groups:
- Placebo + Naive Group: Healthy male and female subjects, aged 22 to 50 years, who previously received placebo in the H03_01TP parent study and who had undetectable antibodies at baseline (Placebo Group), or subjects who were not part of H03_01TP parent study (Naïve Group) were pooled into the Placebo + Naïve Group. All subjects received one intramuscular GVGH Shigella sonnei 1790GAHB vaccine dose in the current study, at Day 1.
Arm/Group | Shigella Group | Placebo + Naive Group
Number analyzed (Participants) | 7 | 28
Participants | 0 | 0

7. Secondary Outcome: Concentrations of IgG Against LPS S. Sonnei O-antigen
Description: Concentrations of IgG against S.sonnei O-antigen are presented as GMCs, expressed in ELISA units per milliliter (EU/mL).
Time Frame: At Days 15, 29 and 85 (14, 28 and 84 days after vaccination)
Population: The analysis was performed on the Full Analysis Set, which included all enrolled subjects who received a study vaccination and who provided immunogenicity data at relevant time points.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Shigella Group | Placebo Group | Naïve Group
Number analyzed (Participants) | 7 | 2 | 25
EU/mL
  Day 15 | 883 [249 to 3126] | 36 [0.89 to 1474] | 106 [53 to 211]
  Day 29: number analyzed (Participants) | 7 | 2 | 24
  Day 29 | 623 [159 to 2446] | 35 [2.36 to 531] | 110 [56 to 213]
  Day 85 | 451 [113 to 1797] | 47 [0.51 to 4250] | 94 [48 to 184]

8. Secondary Outcome: Anti-LPS S. Sonnei IgG Geometric Mean Ratios
Description: Within-subject Geometric mean ratios (GMRs) were computed for GMCs at 7, 14, 28 and 84 days after vaccination versus baseline (Day 1). The GMRs and 95% confidence intervals (CIs) were constructed by exponentiating the mean within-subject differences in log-transformed concentrations and the corresponding 95% CIs.
Time Frame: At Days 8, 15, 29 and 85 (7, 14, 28 and 84 days after vaccination)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Shigella Group | Placebo Group | Naïve Group
Number analyzed (Participants) | 7 | 2 | 25
Ratio
  Day 8/Day 1: number analyzed (Participants) | 7 | 2 | 23
  Day 8/Day 1 | 6.87 [2.69 to 18] | 1.49 [0.0095 to 233] | 2.32 [1.42 to 3.82]
  Day 15/Day 1 | 36 [14 to 93] | 10 [0.26 to 424] | 6.88 [3.77 to 13]
  Day 29/Day 1: number analyzed (Participants) | 7 | 2 | 24
  Day 29/Day 1 | 26 [8.88 to 73] | 10 [0.68 to 153] | 7.21 [4.03 to 13]
  Day 85/Day 1 | 18 [5.37 to 64] | 13 [0.15 to 1223] | 6.11 [3.43 to 11]

9. Secondary Outcome: Percentage of Subjects With Seroresponse for Anti-LPS S. Sonnei
Description: Seroresponse is aimed to define a significant increase in post-vaccination samples based on the biological performance of this specific serology assay and it is defined as follows: - If the baseline value is greater than 50 ELISA Units (EU) then an increase of at least 50% in the post-vaccination sample as compared to baseline [i.e. ((Post-vac minus baseline)/baseline)100% ≥ 50%]. - If the baseline value is less or equal to 50 EU then an increase of at least 25 EU in the post-vaccination sample as compared to baseline [i.e. (Postvac minus baseline) ≥ 25 EU.
Time Frame: At Days 8, 15, 29 and 85 (7, 14, 28 and 84 days after vaccination)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Shigella Group | Placebo Group | Naïve Group
Number analyzed (Participants) | 7 | 2 | 25
Percentage of subjects
  Day 8 | 86 [42.1 to 99.64] | 0 [0 to 84.2] | 26 [10.2 to 48.4]
  Day 15 | 100 [59.0 to 100.0] | 50 [1.3 to 98.7] | 72 [50.6 to 87.9]
  Day 29: number analyzed (Participants) | 7 | 2 | 24
  Day 29 | 100 [59.0 to 100.0] | 100 [15.8 to 100.0] | 67 [44.7 to 84.4]
  Day 85 | 100 [59.0 to 100.0] | 100 [15.8 to 100.0] | 64 [42.5 to 82.0]

10. Secondary Outcome: Percentage of Subjects With Anti-LPS S. Sonnei Concentrations Equal to or Above (≥) 121 EU/mL
Description: Anti-LPS S.sonnei antibody concentrations were assessed by ELISA. The assay cut-off value was 121 EU/mL.
Time Frame: At Days 8, 15, 29 and 85 (7, 14, 28 and 84 days after vaccination)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Shigella Group | Placebo Group | Naïve Group
Number analyzed (Participants) | 7 | 2 | 25
Percentage of subjects
  Day 8: number analyzed (Participants) | 7 | 2 | 23
  Day 8 | 71 [29.0 to 96.3] | 0 [0.0 to 84.2] | 30 [13.2 to 52.9]
  Day 15 | 86 [42.1 to 99.64] | 0 [0.0 to 84.2] | 40 [21.1 to 61.3]
  Day 29: number analyzed (Participants) | 7 | 2 | 24
  Day 29 | 86 [42.1 to 99.64] | 0 [0.0 to 84.2] | 42 [22.1 to 63.4]
  Day 85 | 86 [42.1 to 99.64] | 0 [0.0 to 84.2] | 40 [21.1 to 61.3]

ADVERSE EVENTS:
Time Frame: Solicited local and systemic adverse events: from 30 minutes up to Day 7 post-vaccination; Unsolicited adverse events: throughout the study period (from Day 1 up to Day 85); Serious adverse events: throughout the study period (from Day 1 up to Day 85).
Description: For the purpose of the safety analysis, the subjects from Placebo and Naïve Groups were pooled into a single group (Placebo+Naïve Group). Both groups include vaccine naïve subjects since the placebo recipients in the parent trial did not receive a Shigella vaccine, nor did the naïve subjects who were not part of the parent trial.
Arm/Group | Shigella Group | Placebo + Naïve Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/28
Other Adverse Events (participants affected / at risk) | 7/7 | 25/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Shigella Group (N=7) | Placebo + Naïve Group (N=28)
Chills (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 3 (3) | 11 (12)
Injection site erythema (General disorders) | 2 (2) | 8 (8)
Injection site induration (General disorders) | 2 (2) | 10 (10)
Injection site pain (General disorders) | 6 (6) | 24 (24)
Malaise (General disorders) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (8)
Headache (Nervous system disorders) | 2 (3) | 6 (9)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-02-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT03089879/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-29): https://cdn.clinicaltrials.gov/large-docs/79/NCT03089879/SAP_001.pdf